CLINICAL TRIAL: NCT03498404
Title: Evaluation of Antimicrobial Photodynamic Therapy in Multiple Applications as a Coadjuvant in the Surgical Therapy of Access to Scaling in Patients With Advanced Chronic Periodontitis
Brief Title: Evaluation of Antimicrobial Photodynamic Therapy in Multiple Applications as a Coadjuvant in the Surgical Therapy of Access to Scaling
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Uislen Berian Cadore (Unknown)
Responsible Party: Principal Investigator, Sergio Luis Scombatti de Souza, Dr, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 58437816.3.0000.5419
Record Dates: First submitted 2018-04-07; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Photochemotherapy; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photodynamic Therapy and SRP (Experimental): Procedure/Surgery: Photodynamic Therapy After a surgical access, the periodontal pockets of teeth selected to receive antimicrobial photodynamic therapy (aPDT) will be irrigated with distilled water. Shortly thereafter, the dye will be applied (phenothiazine hydrochloride- 10mg/mL) from the bottom of the pocket. After 1 minute, irrigation will be performed with distilled water to remove the excess of dye. The stained area will be irradiated with a diode laser (660 nm and a 60 mW/cm²). Six sites per tooth under treatment will be irradiated (10 seconds/ site). Teeth with furcation lesion will increase over 60 seconds into the lesion. Before the application, the supragingival plaque will be removed.
  Treatment with TFDa in the Test Group maintained the protocol of applications in the periods of 2, 7 and 14 days post-surgical intervention.
  Interventions: Radiation: Photodynamic Therapy
- SRP and Sham Photodynamic Therapy (Sham Comparator): Procedure/Surgery: Sham Photodynamic Therapy After a surgical access, the periodontal pockets of teeth selected will receive a simulation of antimicrobial photodynamic therapy (aPDT): irrigation with distilled water and simulated laser application. Before the application, the supragingival plaque will be removed.
  Interventions: Other: scaling and root planing

INTERVENTIONS:
Radiation: Photodynamic Therapy — After the sites are indicated for surgical therapy, they receive surgical access therapy associated with scaling and root planing and TfdA using the treatment protocol during periods of 0, 7, 14 and 30 postoperative days, or only surgical access therapy associated with scaling and root planing. As protocol, TfdA will be used laser light source 660nm wavelength in combination with phenothiazine, a photosensitizer with 10 seconds of exposure per site during surgery and 60 seconds in other applications.
  Arms: Photodynamic Therapy and SRP
Other: scaling and root planing — Scaling and root planing, also known as conventional periodontal therapy, or deep cleaning, is a procedure involving removal of dental plaque and calculus (scaling or debridement) and then smoothing, or planing, of the (exposed) surfaces of the roots, removing cementum or dentine that is impregnated with calculus, toxins, or microorganisms, the etiologic agents that cause inflammation. This helps to establish a periodontium that is in remission of periodontal disease. Periodontal scalers and periodontal curettes are some of the tools involved.
  Arms: SRP and Sham Photodynamic Therapy

SUMMARY:
Chronic periodontitis is an infectious disease resulting in inflammation of the teeth support structures, progressive periodontal attachment loss and bone loss. The aim of this study is to evaluate the effects of antimicrobial photodynamic therapy (TFDA) in multiple applications as an adjunct to surgical periodontal therapy in patients with generalized severe chronic periodontitis. A total of twenty patients will be submitted to this split-mouth trial, receiving initial periodontal basic nonsurgical treatment that is scaling and root planing. After the sites are indicated for surgical therapy, they receive surgical access therapy associated with scaling and root planing and TfdA using the treatment protocol during periods of 0, 7, 14 and 30 postoperative days, or only surgical access therapy associated with scaling and root planing. As protocol, TfdA will be used laser light source 660nm wavelength in combination with phenothiazine, a photosensitizer with 10 seconds of exposure per site during surgery and 60 seconds in other applications. All patients will be oral hygiene care and follow-up for 90 days. In the baseline period, basic post-therapy, 30 and 90 days after surgical therapy will be performed the clinical evaluation of plaque index, depth of probing pocket, level of clinical insertion relative and bleeding on probing, beyond the collection plate samples subgingival 40 for counting microbial species using the method of DNA-DNA hybridization checkerboard. For the same periods are also collected samples of gingival crevicular fluid for evaluating fluid volume (Periotron) and the levels of Interleukin 1 beta, Interleukin 10, MMP-8, tumor necrosis factor alpha, RANK-L and Osteoprotegerin (OPG). The data are statistically analyzed with the tests to the sample.

DETAILED DESCRIPTION:
Non-Surgical Periodontal Therapy

Seven days prior to the non-surgical periodontal therapy, periapical radiographs will be taken from the whole mouth of all patients. They will be set in an oral hygiene program (OHP) according to their specific needs. In this program, patients will be instructed about an effective self-performed plaque control, including information about the Bass Technique (Bass, 1954) and interproximal cleaning with dental floss and interdental brushes. They will be also motivated to brush the dorsal surface of the tongue once a day and will receive a dentifrice that shall be used throughout the experimental period (Colgate Total®, Anakol Ind. Com Ltda - Brazil's Kolynos - Colgate Palmolive Co., Sao Bernardo do Campo, SP, Brazil). After the OHP, subjects will undergo the assessment of clinical periodontal parameters previously described and the collection of subgingival plaque and GCF in selected sites (baseline) will be performed. Shortly, patients will receive supragingival scaling and coronal polishing with prophy cup on all the teeth present in the oral cavity. The non-surgical periodontal therapy will initiate 7 days after the OHP and initial supragingival scaling. Within 24 hours, a specialist in Periodontics will perform supra and subgingival scaling and root planing of all teeth with periodontal involvement, using hand (Gracey Curettes, Hu-Friedy, Chicago, IL, USA) and ultrasonic instruments. The instrumentation will be performed on each quadrant until achievement of an adequate cleaning and root planing, which will be verified with a dental explorer. Individuals will receive professional prophylaxis biweekly during three months after the end of the nonsurgical periodontal therapy. On biweekly follow-up visits, patient's cooperation will be monitored by verifying the status of oral hygiene.

Surgical Periodontal Therapy

The flap operations are performed 8 weeks after the start of the basic preparation. Patients will be monitored clinically and sites that present PS ≥ 5mm and SS presence will undergo surgical therapy scraping retail. Surgical procedures will be performed by a specialist in Periodontics. Initially patients will be subjected to extra-oral antisepsis with chlorhexidine 2% and intraoral through mouthwash with chlorhexidine 0.12%. The region to be operated infiltrative receive local anesthesia with lidocaine 2% solution, and 1: 100,000 epinephrine. The following will be performed intra-sulcular incision with a scalpel blade at 15C covering the site with PS ≥ 5mm and the adjacent teeth. A mucoperiosteal flap will be performed until the exposure of the bone crest and subgingival deposits of calculation and / or granulation tissue are removed by conventional Gracey curettes with RAR and Mini Five, numbers 5/6, 7/8, and 11/12 13/14 (Hu-Friedy, Chicago, IL, USA) and ultrasonic devices. Shortly after completion of the RAR starts to tfdA the operated region in the selected adjuvant therapy for this group. Completed therapy, the flap will be positioned in the same place of origin and stabilized with simple sutures through wire Vicryl 5-0. In order to avoid painful symptoms will be prescribed analgesics (Paracetamol 750mg, 01 tablet every 6 hours for 48 hours). They will also be prescribed soft oral rinses with 0.12% chlorhexidine digluconate, 2 times a day for 14 days. The sutures are removed after 7 days. Being performed weekly supragingival plaque control in the first month and monthly until completing 3 after surgical intervention months.

Antimicrobial photodynamic Therapy

After surgical access and realization of flap RARÎ, surgical sites selected to receive the TfdA will be irrigated with saline will be dried with sterile gauze, a period of 10 minutes and waited, until there is no more bleeding. Soon after, will be applied fotossintentizador hydrochloride phenothiazine, whose main component is the toluidine blue at a concentration of 10mg / mL (Helbo Blue, Helbo Photodynamic Sytems, Grieskirchen, Austria), which will be in contact for 3 minutes. Posteriorly, irrigation will be performed with saline solution for removal of the excess fotossensitizador and colored areas are irradiated with a laser diode of wavelength 660 nm, maximum power 60 mW / cm2 and an energy density of 0,6J / cm2 ( Helbo therapielaser, Helbo Photodynamic Systems GmbH & Co KG, Grieskirchen, Austria), for 60 seconds per site. The treatment is carried out in 6 sites on the teeth, totaling six minutes of application of laser light per tooth. Teeth with furcation lesion will increase more 60 seconds into the lesion.

Each patient will be impressed with alginate in order to obtain models of the dental arches and elaborate a guide plate made of acetate. This plate will present grooves that will be used as references to standardize the insertion and tilt of the automated periodontal probe (Florida Probe System, Florida Probe Corporation, Gainesville, FL, USA). The visible plaque index for each patient, rated dichotomously (O'Leary et al. 1972), will be determined by the percentage of tooth surfaces with deposits of plaque stained with disclosing solution.

Post-surgical protocol

Treatment with TFDa in the Test Group maintained the protocol of applications in the periods of 2, 7 and 14 days post-surgical intervention as described by (Ramos et al., 2016). This protocol is distinct from the previous one by the time of exposure to laser light. In the protocol described above, the exposure time is 60 seconds per site totaling 6 minutes. In this, the applications are only 10 seconds per site at 6 sites per tooth, totaling 1 minute of exposure. Teeth involving bifurcation lesion had an additional 10 seconds inside the lesion.

Clinical monitoring

The following clinical periodontal parameters will be assessed at 6 sites of each tooth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual and disto-lingual): (i) probing pocket depth (PPD): it will be measured from the gingival margin to the bottom of the pocket; (ii) gingival recession (GR): it will be measured from the enamelcement junction to the bottom of the pocket; (iii) clinical attachment level (CAL): it will be measured as PPD + GR (GR will be equal to 0 whenever the cementenamel junction is covered); (iv) bleeding on probing (BOP): it will be evaluated dichotomously: the presence of the bleeding will be considered positive when occurring within 30 seconds from the insertion of the probe for probing depth; (v) Plaque index (PI): it will be evaluated dichotomously. BOP, PPD, CAL and GR will be measured at six sites per tooth (mesio-buccal, buccal, disto-buccal, disto-lingual, lingual and mesio-lingual). All probing measurements will be performed using an automated periodontal probe.

The clinical periodontal parameters and the plaque index of each patient will be recorded at baseline (pre-intervention), as well as +30 and +90 days after the surgical periodontal therapy. The Kappa index will be used to evaluate the examiner calibration on clinical periodontal parameters collection in order to calculate the intra-examiner agreement. According to the World Health Organization (WHO) criteria for diagnosis, the acceptable Kappa index of agreement must be greater than or equal to 0.85 (WHO, 1997). This level of agreement will be used for calibration of the examiner in this project. Ten patients, each one showing at least two pairs of contralateral single-rooted teeth with PD ≥ 5 mm on interproximal sites, will be selected to calibrate the examiner. Each patient will be evaluated on two separate occasions 48 hours apart in order to obtain the intra-examiner reliability through the Kappa index.

Microbiological monitoring

At baseline and +30 and +90 days after the surgical periodontal therapy, samples of subgingival plaque will be obtained from eight interproximal sites of each patient. Samples will be individually analyzed for their content of 40 subgingival bacterial species using the checkerboard DNA-DNA hybridization technique (Socransky et al., 2004a; Socransky et al., 2004b). The selected teeth will be isolated with sterile cotton rolls and dried with air jets. Then, the supragingival plaque will be carefully removed using a sterile curette. Another sterile curette will be used to collect the subgingival plaque, starting from the bottom of the periodontal pocket to its coronal portion. The samples will be stored in sterilized Eppendorf tubes and will be processed at the Microbiology Laboratory of the Guarulhos University (UNG, Guarulhos, SP, Brazil).

Statistical analysis

The normality and homoscedasticity of the data obtained will be checked. Comparisons within groups and among groups at different time intervals will be performed through parametric or non-parametric appropriate tests. The significance level will be set at 5% in all tests. All calculations will be performed by SPSS software (SPSS, Chicago IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with >35 years old
* A minimum of 15 teeth present
* One pair of posterior teeth in opposite sides with proximal sites showing probing depth and clinical attachment level ≥ 5 mm.

Exclusion Criteria:

* Positive history of antibiotic-therapy in the last six months
* Positive history of basic periodontal treatment in the last six months
* Systemic disease that can interfere with the progression of disease or response to treatment (eg, diabetes, immune disorders)
* Extensive prosthetic involvement
* Need for antibiotic prophylaxis for performing routine dental procedures
* Use of anti-inflammatory drugs for long periods of time
* Smoking
* Pregnancy

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-07 (Actual); Primary Completion 2018-04-07 (Actual); Study Completion 2018-04-07 (Actual)

PRIMARY OUTCOMES:
to evaluate clinical attachment level | The clinical periodontal parameter will be recorded at baseline (pre-intervention) and +120 days after the surgical periodontal therapy.
  Change from Baseline in clinical attachment level at +120 days

SECONDARY OUTCOMES:
counts of 40 subgingival bacterial species | Microbiological monitoring (at baseline and +30 and +120 days after the surgical periodontal therapy) using the checkerboard DNA-DNA hybridization
  Change from baseline in counts of 40 subgingival bacterial species at +30 and +120 days
patients requiring additional periodontal treatment | Considering each group separately, it will be evaluate the number of patients presenting at least a site with PPD≥5 mm and positiveBOP at 120 days post-therapy
  Numbers of patients requiring additional periodontal treatment at +120 days.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided